CLINICAL TRIAL: NCT03335436
Title: A Randomized, Double-blind, Placebo-controlled Trial of Gabapentin in the Post-cesarean Pain Management of Buprenorphine Patient
Brief Title: Gabapentin in the Post-cesarean Pain Management of Buprenorphine Patient
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Holly Ende, Asst Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 171688
Record Dates: First submitted 2017-10-09; First posted 2017-11-07 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Cesarean Delivery; Pain Management
Keywords: buprenorphine maintenance
MeSH Terms: conditions — Agnosia | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gabapentin (Experimental): Gabapentin 600 mg by mouth one hour prior to scheduled cesarean delivery and 400 mg by mouth every 8 hours post delivery
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): Placebo with similar appearance to gabapentin by mouth one hour prior to scheduled cesarean delivery and by mouth every 8 hours post delivery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Participants will receive Gabapentin 600 mg by mouth one hour prior to scheduled cesarean delivery and 400 mg by mouth every 8 hours post delivery
  Arms: Gabapentin
Drug: Placebo — Participants will receive Placebo with similar appearance to gabapentin by mouth one hour prior to scheduled cesarean delivery and by mouth every 8 hours post delivery
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether a perioperative course of gabapentin in parturients on buprenorphine maintenance would improve analgesia after elective cesarean delivery (CD).

DETAILED DESCRIPTION:
Many strategies have been suggested to improve post-CD pain management in parturients on buprenorphine. While effective pain relief can be achieved, women maintained on buprenorphine during pregnancy have been shown to require up to 50% more opioids after CD compared to women with opioid use disorder not on a maintenance regimen. The perioperative use of gabapentin has been shown to reduce pain scores and opioid consumption following a variety of surgeries, ranging from cardiac bypass to total abdominal hysterectomy. The purpose of this study is to determine whether a perioperative course of gabapentin in parturients on buprenorphine maintenance would improve analgesia after elective CD.

ELIGIBILITY:
Inclusion Criteria:

* singleton, term pregnancy
* currently on buprenorphine maintenance therapy
* scheduled for elective CD under spinal anesthesia

Exclusion Criteria:

* use illicit drugs or relapse during the last trimester of pregnancy
* positive drug screen at the time of delivery
* allergies to any medications used in the study
* taking prescribed gabapentin at the time of admission for CD
* contraindications to neuraxial anesthesia or require general anesthesia for CD
* designated ASA physical status 4 or above

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Total opioid use 24 hours after cesarean delivery | 24 hours after cesarean delivery
  Total opioid use tallied in morphine milligram equivalents at 24 hours after cesarean delivery
Total opioid use at time of hospital discharge after cesarean delivery | From the end of cesarean delivery to the time of hospital discharge after cesarean delivery, approximately 4 days
  Total opioid use tallied in morphine milligram equivalents from the end cesarean delivery to the time of hospital discharge after cesarean delivery

SECONDARY OUTCOMES:
Pain assessment using 11-point Visual/Verbal Analog (VAS) at rest 4 hours post-partum | 4 hours post-partum
  Pain assessment using VAS at rest 4 hours post-partum when 0 is no pain and 10 is worst pain
Pain assessment using 11-point Visual/Verbal Analog (VAS) at movement 4 hours post-partum | 4 hours post-partum
  Pain assessment using VAS at movement 4 hours post-partum when 0 is no pain and 10 is worst pain
Pain assessment using 11-point Visual/Verbal Analog (VAS) at rest 24 hours post-partum | 24 hours post-partum
  Pain assessment using VAS at rest 24 hours post-partum when 0 is no pain and 10 is worst pain
Pain assessment using 11-point Visual/Verbal Analog (VAS) at movement 24 hours post-partum | 24 hours post-partum
  Pain assessment using VAS at movement 24 hours post-partum when 0 is no pain and 10 is worst pain
Pain assessment using 11-point Visual/Verbal Analog (VAS) at rest 48 hours post-partum | 48 hours post-partum
  Pain assessment using VAS at rest 48 hours post-partum when 0 is no pain and 10 is worst pain
Pain assessment using 11-point Visual/Verbal Analog (VAS) at movement 48 hours post-partum | 48 hours post-partum
  Pain assessment using VAS at movement 48 hours post-partum when 0 is no pain and 10 is worst pain
Pain assessment using 11-point Visual/Verbal Analog (VAS) at rest 30 days post-partum | 30 days post-partum
  Pain assessment using VAS at rest 30 days post-partum when 0 is no pain and 10 is worst pain
Pain assessment using 11-point Visual/Verbal Analog (VAS) at movement 30 days post-partum | 30 days post-partum
  Pain assessment using VAS at movement 30 days post-partum when 0 is no pain and 10 is worst pain
Presence of persistent pain | 30 days post-partum
  Presence of persistent pain defined as pain score greater than baseline at 30 days post-partum
Return to normal daily function | 30 days post-partum
  Return to normal daily function assessed with the Veterans RAND 12-item questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Holly B Ende, M.D,, Principal Investigator — Vanderbilt University Medical Center

IPD SHARING:
Plan to Share IPD: No